CLINICAL TRIAL: NCT04893967
Title: Effects of Magnetic Tape on Isometric Hip Strength in Patients With Low Back Pain. RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clínica Dr. Francisco Selva (Other)
Responsible Party: Principal Investigator, Francisco Selva, Director PhD, Clínica Dr. Francisco Selva
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1622496
Record Dates: First submitted 2021-05-10; First posted 2021-05-20 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2021-05

CONDITIONS: Low Back Pain
Keywords: strength; pain; low back pain; dynamometer; abduction; surface electromyogram; magnetic tape; kinesiology tape; Hip Stability Isometric Test (HipSIT)
MeSH Terms: conditions — Low Back Pain; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (18):
- No Intervention: RMS mean hip abduction, dynamometer (No Intervention): Isometric peak force hip abduction pre measurement. No tape.
- No Intervention: Average force hip abduction, dynamometer (No Intervention): Isometric average force hip abduction pre measurement. No tape.
- No Intervention: Time to reach peak force hip abduction, dynamometer (No Intervention): Time to reach peak force hip abduction pre measurement. No tape.
- No Intervention: RMS mean hip abduction, surface electromyogram (No Intervention): Isometric hip abduction pre measurement assessing the root-mean-square (RMS) mean. No tape.
- No Intervention: RMS mean per second hip abduction, surface electromyogram (No Intervention): Isometric hip abduction pre measurement assessing the root-mean-square (RMS) mean per second. No tape.
- No Intervention: Max. contraction test hip abduction, surface electromyogram (No Intervention): Isometric hip abduction pre measurement assessing the root-mean-square (RMS) Max. contraction test. No tape.
- Experimental: peak force hip abduction, dynamometer (Experimental): Isometric peak force hip abduction post experimental application measurement with Magnetic Tape application
  Interventions: Device: Magnetic Tape
- Experimental: Average force hip abduction, dynamometer (Experimental): Isometric average force hip abduction post experimental application measurement with Magnetic Tape application
  Interventions: Device: Magnetic Tape
- Experimental: time to maximum force hip abduction, dynamometer (Experimental): Time to maximum force hip abduction post experimental application measurement with Magnetic Tape application
  Interventions: Device: Magnetic Tape
- Experimental: RMS mean hip abduction, surface electromyogram (Experimental): Isometric hip abduction post experimental application measurement assessing the root-mean-square (RMS) with Magnetic Tape application.
  Interventions: Device: Magnetic Tape
- Experimental: RMS mean per second hip abduction, surface electromyogram (Experimental): Isometric hip abduction post experimental application measurement assessing the root-mean-square (RMS) mean per second. With Magnetic Tape application.
  Interventions: Device: Magnetic Tape
- Experimental: Max. contraction test hip abduction, surface electromyogram (Experimental): Isometric hip abduction post experimental application measurement assessing the root-mean-square (RMS) max. contraction test. With Magnetic Tape application.
  Interventions: Device: Magnetic Tape
- Placebo: peak force hip abduction, dynamometer (Placebo Comparator): Isometric peak force hip abduction post placebo measurement with kinesiology tape application
  Interventions: Device: kinesiology tape
- Placebo: Average force hip abduction, dynamometer (Placebo Comparator): Isometric average force hip abduction post placebo application measurement with kinesiology tape application
  Interventions: Device: kinesiology tape
- Placebo: Time to reach peak force hip abduction, dynamometer (Placebo Comparator): Time to reach peak force hip abduction post placebo application measurement with kinesiology tape application
  Interventions: Device: kinesiology tape
- Placebo: RMS mean hip abduction, surface electromyogram (Placebo Comparator): Isometric hip abduction post placebo application measurement assessing the root-mean-square (RMS) mean. With kinesiology tape application.
  Interventions: Device: kinesiology tape
- Placebo: RMS mean per second hip abduction, surface electromyogram (Placebo Comparator): Isometric hip abduction post placebo application measurement assessing the root-mean-square (RMS) mean per second. With kinesiology tape application.
  Interventions: Device: kinesiology tape
- Placebo: Max. contraction test hip abduction, surface electromyogram (Placebo Comparator): Isometric hip abduction post placebo application measurement assessing the root-mean-square (RMS) max. contraction test. With kinesiology tape application.
  Interventions: Device: kinesiology tape

INTERVENTIONS:
Device: Magnetic Tape — Magnetic tape® is applied without creating any tension over low back
  Arms: Experimental: Average force hip abduction, dynamometer; Experimental: Max. contraction test hip abduction, surface electromyogram; Experimental: RMS mean hip abduction, surface electromyogram; Experimental: RMS mean per second hip abduction, surface electromyogram; Experimental: peak force hip abduction, dynamometer; Experimental: time to maximum force hip abduction, dynamometer
Device: kinesiology tape — Kinesiology Tape is applied without creating any tension over low back
  Arms: Placebo: Average force hip abduction, dynamometer; Placebo: Max. contraction test hip abduction, surface electromyogram; Placebo: RMS mean hip abduction, surface electromyogram; Placebo: RMS mean per second hip abduction, surface electromyogram; Placebo: Time to reach peak force hip abduction, dynamometer; Placebo: peak force hip abduction, dynamometer

SUMMARY:
The tape will be applied on the lumbar area bilaterally to the spine without creating any tension.

The possible variation in the isometric hip strength is measured with the mDurance®, surface electromyography and the Lafayette® dynamometer. A kinesiology tape was used as a placebo tape and the magnetic tape was used in a randomized experimental way.

DETAILED DESCRIPTION:
A doble-blind clinical trial study, is designed where subjects with low back pain will be selected and blinded to receive the Magnetic Tape® or placebo Tape. Likewise, the evaluator who puts the Magnetic Tape® does not know what material he is using, as it is supplied by another researcher. The patient does not know what tape will be placed on him.

The recommendations of the "Consolidated Standards of Reporting Trials" (CONSORT) will be followed. All participants will receive a participant information sheet and sign informed consent. Patients aged 18 to 65 years with low back pain will be recruited from different private clinics in the city of Valencia, Spain.

The hypothesis is that when Magnetic Tape® comes into contact with electromagnetic fields such as those generated by living beings, due to the movement of electrical charges (ions), as defined by Ampere's Law, the domains of the tape are oriented or aligned in parallel with the external magnetic field creating a magnetic flux with a north pole and a south pole. This generated field in turn produces a magnetic induction proportional to the variation of the magnetic flux, as defined by the Faraday Law.

This electric potential produces a redistribution of the electric charge (ions) generating a magnetic field due to the orientation of the tape domains, then exerting a force on the moving charges within the electrolyte.

Physiological, Lorentz's Law, regulating Magnetic Tape® aberrant electromagnetic fields.

The protocol for data collection will be as follows:

After signing the informed consent and data protection, the groups with low back pain will be formed that will receive the application of both Magnetic Tape® and the intervention of a placebo tape. To avoid that the order of the intervention influences the results of the study, the subjects will be randomized into two different groups, Group A and Group B. Group A will receive Magnetic tape® and Group B will do the opposite. The next day the other tape.

To evaluate the isometric force of hip abduction or Hip Stability Isometric Test (HipSIT). A surface electromyogram and a force dynamometer are used. The electrodes of the surface electromyogram will be placed on the Tensor Fascia Lata and Gluteus Medius muscles bilaterally. The patient will be placed in lateral decubitus with 45 ° hip flexion and 90 ° knees. Both lower limbs will be cinched over the distal third of the thigh where the center of the Lafayette dynamometer will be positioned laterally 5 cm above the knee joint. The subject will perform the separation of the upper hip while keeping the heels in contact so that the hip is in 20 ° of abduction, using its maximum force for 5 seconds performing it 4 times resting between tests for 30 seconds and recording the electromyographic activity.

The tapes will be placed on the paravertebral skin from L1 to L5 without creating tension.

Subsequently, both hips are assessed again, performing hip abduction again and recording the strength.

Each subject will be your control since one day a tape will be placed and the next day the other.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with low back pain.
* Subjects aged 18-65 years.

Exclusion Criteria:

* Tape allergies
* Adhesive allergies
* Pregnant
* People with pacemakers
* People who have any contraindication of electromagnetic fields
* People with neurological diseases
* Taking any medication that may interact with magnetic fields.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
muscle fiber activation | Changes for activity (microvolts) first evaluation before placing the tapes and immediately after placing the experimental tape and the placebo tape.
  Maximum isometric strength of hip abduction measured with the mDurance® surface electromyograph.
Peak force of hip abduction | Changes from strength (kilograms) in first assessment before placing the tapes and immediately after placing experimental tape and placebo tape.
  Maximum isometric strength of hip abduction measured with the Lafayette® dynamometer.
Average force of hip abduction | Changes from strength (kilograms) in first assessment before placing the tapes and immediately after placing experimental tape and placebo tape.
  Mean isometric strength of hip abduction measured with the Lafayette® dynamometer.
Time to reach peak force of hip abduction | Changes from time (seconds) in first assessment before placing the tapes and immediately after placing experimental tape and placebo tape.
  Time to maximum isometric strength of hip abduction measured with the Lafayette® dynamometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Francisco Selva, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No